CLINICAL TRIAL: NCT00388921
Title: High/Low Dose Vit A in Diarrhea/ALRI in Severe PEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-033
Record Dates: First submitted 2006-10-15; First posted 2006-10-17 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2005-11

CONDITIONS: Respiratory Infections; Diarrhea; Malnutrition
Keywords: Vitamin A; Children; Severe malnutrition; Retinol; Retinol binding protein; Diarrhoea; ALRI; Age 6-59 months; Either sex; Severe malnutrition as defined by the presence of any of the followings:; Bipedal oedema; Weight (measured after correction of dehydration) for height Z score <-3 of the National Center for Health Statistics (NCHS) reference; Written informed consent of respective parents/ guardians for participation of the children in the study.; Children having diarrhoea (watery or invasive) or cough and cold or both for the last 48 hours.
MeSH Terms: conditions — Respiratory Tract Infections; Diarrhea; Malnutrition; Body Weight; Cough; Common Cold | interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
Vitamin A deficiency is an important health problem globally including Bangladesh. The problem is greater among under-five children, particularly in malnourished. Vitamin A supplementation reduces morbidity from diarrhoeal diseases and also prevents future diarrhoea episodes. However, there are conflicting reports on the role of vitamin A supplementation on morbidity from acute lower respiratory infections (ALRI) including pneumonia. In non-malnourished children supplementation has been reported to be associated with increased incidence and morbidity of ALRI. The WHO committee[1] has reviewed both the risk and benefit of mega dose (200,000 IU) vitamin A supplementation during acute illness particularly diarrhoea, irrespective of the nutritional status of under-5 children and recommended vitamin A supplementation in areas where vitamin A status is low. In Bangladesh mega dose (200,000 IU) of vitamin A is routinely supplemented to under-5 children every 6 months. Absorption of vitamin A precursors from the GI tract is reduced in severely malnourished children, who are also lacking in retinol binding protein (RBP), required for transportation of retinol to target tissues. Thus it is established that a significant portion of the supplemented vitamin A is excreted in feces and urine of malnourished children. The excretion of vitamin A increases substantially during acute infections including diarrhoeal diseases. On the other hand, due to reduced RBP, concentration of free vitamin A increases in the body resulting in the possibility of adverse events including "pseudotumor cerebri". It has recently been observed that low-dose daily supplementation of vitamin A to malnourished children produces a better effect on recovery from acute illness and also in preventing infectious diseases among under-five children. However, the limitations of those studies included a small sample size, delayed assessment of retinol after supplementation among the others. Thus WHO felt that the issue needs to be addressed in a well-designed clinical trial. We hope that our proposed study will enable us to compare the efficacy of low-dose daily administration of vitamin A with that of initial mega dose followed by daily low dose of vitamin A in malnourished children presenting with acute diarrhoeal diseases with or without ALRI. If the results of this study indicate that the daily low-dose has similar efficacy to that of the currently recommended mega dose followed by daily low-dose of vitamin A, would have important programmatic implications.

DETAILED DESCRIPTION:
Globally An estimated 140-250 million under-five children are deficient in vitamin A, which is associated with increased mortality and morbidity among this population. A relationship between the severity of vitamin A deficiency and childhood mortality has also been reported. In 2002, the United Nations held a special session to examine ways to eliminate this problem through various approaches including breast-feeding, food fortification, improved diet and supplementation. Periodic supplementation of a mega dose of vitamin A has been recommended to be a suitable intervention at the community level which is likely to improve the over all vitamin A status. This is also cost effective and patient compliant. This approach has resulted in reduction in all-causes of deaths among under-five children by 23% in areas where vitamin A deficiency is a major public health problem [3] (http://www.who.int/vaccines/en/vitamina.shtml accessed on 26 May, 2005 at 1300 hrs). In view of the public health importance of vitamin A nutriture, the Government of Bangladesh recommends the administration of 200,000 IU of vitamin A every six months to all children aged 12-59 months irrespective of their nutritional and vitamin A status (Institute of Public Health Nutrition. Field guide for National Vitamin A Plus Campaign, 2005).

Vitamin A is required for maintenance of integrity of epithelial cells and its growth and differentiation, visual function, and the immune system [4]. Vitamin A deficiency leads to patchy keratinization of epithelial lining of the respiratory, genitourinary and gastrointestinal tracts [5], which acts as protective barriers against infections. The loss of intestinal epithelial integrity increases the likelihood of bacterial colonization and incidence of infections and septicemia, and it has also been shown that vitamin A supplementation in smaller or higher doses help repair the damaged mucosa during the convalescence stage [6-10]. Vitamin A deficiency state is worsened during acute infections that reduces the dietary intake and absorption, and increases excretion of vitamin A in urine [11]. The mortality in vitamin A deficiency is also related to reduced immune function [12], [13]. Vitamin A improves wound healing by mediating early inflammatory responses associated with influx of macrophages, enhanced fibroblast differentiation, and collagen accumulation [14].

About half of the absorbed vitamin A ingested is oxidized and excreted in the feces and urine, and the remainder is stored in the liver as retinol ester. It is released into the plasma for transportation to peripheral tissues after binding with specific protein known as retinol binding protein (RBP). Protein deficiency in severe malnutrition reduces the hepatic synthesis of RBP [15], [16] which is the likely to be the reason for low serum retinol level observed in such children [17-19]. Infectious diseases such as diarrhoea and acute lower respiratory infections including pneumonia are common in malnourished children, which worsen the vitamin A level [20]. Acute infections are also associated with acute phase response and a transient decrease in serum retinol level [21]. This is due to reduced transcription of messenger RNA for RBP, resulting in decreased release of RBP from the liver into the blood [22], [23]. It is likely that liver utilizes all of its available resources for rapid synthesis of proteins that are required for the host defense in acute infection, thereby limiting the synthesis of relatively lesser important ones such as RBP. In severe infection, the increased urinary loss of retinol contributes to the lower serum retinol concentration [24]. Thus the utilization of vitamin A in the peripheral tissue is adversely affected in systemic infections and in protein- energy malnutrition leading to development of features of vitamin A deficiency.

Acute lower respiratory infections (ALRI) including pneumonia, and diarrhoeal diseases are the two most common illnesses that affect the under-five children. Earlier studies have observed beneficial role of high dose vitamin A as an adjunct therapy in the treatment of both watery and invasive diarrhoeas [25, 26]. It was observed that an increase of 1 mmol/liter of retinol reduces proportion of patients with diarrhoea and respiratory disease by 50% and 80% respectively [9]. A more recent study had observed supplementation of vitamin A to under-five children to be associated with reduced frequency of diarrhoea and ALRI, and subsequent malnutrition [27]. In another study 85% of the infants attending a diarrhoea treatment centre in Bangladesh were found to have depleted vitamin A stores, as measured by relative dose response test, and 61% of them remained deficient despite receiving high dose of vitamin A [24, 28]. Healthy children receiving high dose of vitamin A may experience higher incidences of adverse manifestations such as nausea, vomiting and higher incidence of diarrhoeal episode [29], while low dose vitamin A is associated with reduced incidence of severe diarrhoea in malnourished children [15]. In India studies examined the effect of an intermediate dose (8.7 mmol; 2500 mgm), administered weekly, and did not observe any difference in the incidence, severity and or duration of diarrhea in vitamin A deficient children [30]. In another community based study, infants aged 2-15 months receiving 16700 IU vitamin A or placebo weekly for 8 weeks experienced enhanced gut repair as indicated by improved lactulose-mannitol (L:M) ratio, as compared to the hospitalized infants who received high dose. The results suggest impaired gut permeability during convalescent period. There is every possibility that the low vitamin A level during the infectious state and the low retinol concentration in malnourished children aggravates the already existing compromised gut mucosa thus necessitating the vitamin A supplementation among the hospitalized malnourished children [10].

There are conflicting reports on the role of high dose of vitamin A supplementation in the management of ALRI and pneumonia in malnourished children [31], [15]. Even sub-clinical vitamin A deficiency in non-malnourished children is associated with increased risk of ARI [32], [33]. Meta-analysis of community-based studies of high dose vitamin A supplementation to children aged 6 months to 5 years did not observe any protective or detrimental effects of vitamin A supplementation on pneumonia-specific mortality according to the vitamin A and pneumonia working group [34]. In fact, some studies have reported an increase in the incidence of ALRI in children with adequate nutritional status receiving vitamin A supplementation [35]. In a placebo-controlled study, high dose vitamin A supplementation did neither influence recovery nor the duration of hospitalization in Guatemalan children with ALRI [31]. A higher dose of vitamin A was evaluated in studies in Brazil [36], Vietnam [37], Chile [38] and Tanzania [39], and none of them had observed any beneficial effect, and in fact had observed a negative effect in adequately nourished children [40]. Another clinical trial conducted in Peru not only observed high dose vitamin A supplements to be ineffective in improving recovery from pneumonia in hospitalized children, but actually observed prolonged duration of the clinical signs, higher requirements of oxygen support, and higher nursing time and patient care cost in high-dose supplemented group [41]. On the other hand, in a population based, controlled clinical trial in Ecuadorian urban slum children, weekly supplementation of low dose vitamin A (10,000 IU) for 40 weeks was associated with a strong protective effect on ALRI in malnourished under-five children [42].

The reports on mortality and morbidity from diarrhoea and pneumonia in severely malnourished children in association with vitamin A supplementation are conflicting. In the 21st IVACG meeting three papers were reviewed. They observed no significant difference in mortality (8% vs. 8.4% and 8.8%) in high and low dose of vitamin A and placebo group [15]. Yet another study also failed to show any significant reduction (16.8 vs. 12.4%) in the mortality in patients receiving high or low dose of vitamin A [43]. However, in sub-group analysis deaths were significantly lower among oedematous children who received low dose vitamin A on admission [44]. A meta-analysis observed substantial reduction in mortality in association with vitamin A supplementation in population where at least low-level deficiency state was prevalent, and the effect was independent of dose, sex and age, and the effect was more pronounced for incidence of diarrhoea than for respiratory diseases [45]. However, no difference in morbidity (frequency, duration, or prevalence) from diarrhoeal or respiratory diseases was noted (Ghana VAST Study Team) [46] among stunted children in Ghana.

Malnourished children are deficient in RBP, facilitating excretion of the resultant free, unbound form of vitamin A either through urine or faces, a situation that is aggravated during acute infections. Vitamin A, when administered in a single high dose, presumably circulates in free form in the extra cellular fluids before being taken up by the liver. This free form of vitamin A perhaps affects sodium and water metabolism causing 'pseudotumor cerebri', an adverse event of hypervitaminosis A [47]. Thus a mega dose supplementation may not be yielding any better effect in the severely malnourished children.

Rationale

Vitamin A supplementation is beneficial in the management of clinical and sub-clinical deficiencies of this important micronutrient, and has been observed to improve outcomes from certain illnesses, particularly diarrhoeal diseases and in preventing infectious diseases. The beneficial effect of vitamin A supplementation in ALRI including pneumonia is not that clear. WHO currently recommends single high dose of vitamin A supplementation to malnourished children with diarrhoea because of low cost with high participation rate for improving health status of children. The WHO recommendation is based on studies in communities that showed benefit of the cheapest intervention, which is quicker to implement into health programmes. The programmes for vitamin A capsule distribution reduced risk of vitamin A deficiency among participating children. Interpretation of the three studies done in the Democratic Republic of Congo and Senegal, as mentioned earlier, in relation to the existing guidelines on vitamin A supplementation was considered difficult and their validity was doubted in a meeting convened by WHO in September 2004. It was, however, recognized that the question of vitamin A dosage remains an important one and there is scope for further research. The meeting proposed that the high dose only be given if the interval is at least 6 months from the last previous high dose.

In Bangladesh, high potency (200,000 IU) vitamin A is routinely supplemented to under-five children every 6 months. There are at least three large studies that failed to observe any effect of mega dose of vitamin A on the incidences and duration of diarrhoea and respiratory tract infections. In recent studies it has been shown that daily low-dose supplementation of vitamin A to malnourished under-five children produces similar or better effect, compared to high dose, during acute illness and also in preventing infectious diseases. Studies have observed higher mortality in high dose vitamin A supplemented group compared to the low dose group. However, they were done in smaller number of children [15, 44]. In serum, vitamin A remains saturated with RBP in a 1:1 ratio. Therefore, the amount of vitamin A in excess of this ratio, as would be expected in mega-dose supplementation of vitamin A to severely malnourished children with low serum RBP, would be non-functional at best, at least theoretically [19]. Two trials in Asia that used high dose vitamin A observed conflicting results. One study reported that, capsule distribution was not universal and probably vitamin A deficient children would be missed, and the response of the high dose was unlikely to be due to non-specific changes. In the other study, vitamin A supplementation alone failed to show any expected improvement of child survival in demographic data but they did not deny the importance of vitamin A supplementation in improving nutritional status [48, 49]. On the other hand, weekly supplement of 8,333 IU of vitamin A was reported to reduce mortality by 54% [50]. There thus is a need for a carefully designed study with adequate sample size to address the effect of low dose vitamin A on morbidity and mortality among severely malnourished children with diarrhoea and pneumonia- the basis of our proposed study. We hope that the results of this study will enable us to compare the cure rates of low-dose daily administration of vitamin A with that of the initial mega dose followed by daily low dose of vitamin A. Daily basal requirements (estimated amount which is needed to prevent signs of deficiency) for 0-1 and 2-6 years old children are 600 and 650 IU respectively, and the normal requirement (which is sufficient to maintain desirable levels of tissue store) for the same age group are 1200 and 1300 IU respectively [51]. It is estimated that malnourished children will lose 0.1µmol of retinol /day (97 IU) through urine during acute illness [24].

The national coverage rate (percentage of target age children who received vitamin A capsules during the past six months, according to information provided by the mothers) of vitamin A in rural areas was 45% in 1982-83[52]. The rate gradually decreased to 37% in 1987-88 and 35% in 1989 respectively [53], [54]. However, the Nutritional Surveillance Project reported in December 1995, that the coverage of vitamin A capsule distribution increased substantially- 83.6% in rural and 73.7% in the urban areas [54]. It is noteworthy that night blindness is considered as the marker of vitamin A deficiency, and when that exceeds 1%, is considered as a significant public health problem [55]. In Bangladesh, the proportion of children aged 18-59 months having night blindness in rural areas and urban slums were 0.23% and 0.12% respectively [52]. These figures are well below the cut-off for public health significance of vitamin A deficiency. Anecdotal observations of doctors working at the ICDDR, B Hospital, Dhaka, indicate a significant decrease in the number of children with clinical vitamin A deficiency seeking treatment in the hospital. Further more, according to a report of the surveillance system of Dhaka Hospital of ICDDR, B 84 children presented with conjunctival xerosis and only three had keratomalacia/corneal ulcer out of the total of 11,605 under-5 children who attended the hospital during the period 1996-2004. Children to be enrolled in our proposed study will receive 5000 IU of vitamin A. That amounts to be an additional 1000 IU during the acute phase and 800 IU during the nutritional rehabilitation phase of severe malnutrition from various diets provided to them during their hospital stay. We thus estimate that the total amount of vitamin A received from these sources, even after adjusting for urinary excretion and the retinol level, will not fall below the basal and normal requirements. We feel that once we are able to maintain the daily optimal level of vitamin A stores in the body the sudden development of keratomalacia can be averted. However, we will remain vigilant, through performing careful clinical examination (of eye and skin), to exclude children with any form of clinical vitamin A deficiency from enrollment. Children with clinical vitamin A deficiency disease (conjunctival xerosis, Bitot's spots, keratomalacia, or dermatosis suggestive of vitamin A deficiency) will not be eligible for enrollment and will be provided with the currently recommended treatment with vitamin A supplementation as is routinely followed in this hospital. It may also be noted that a couple of studies did not observe development of an overt sign of vitamin A deficiency in children not receiving vitamin A (placebo group) [15, 41]. Additionally, serum retinol concentrations were not significantly changed after 7 days of hospitalization both among children receiving the high dose and children receiving the low dose or placebo [15].

Clinical failure rates in the first 48 hours for the Dhaka hospital for shigellosis, cholera and pneumonia were 31%, 35% and 40% respectively. Thus we postulate that the clinical failure from diarrhoea and pneumonia will be reduced at least by 15% from the current rate, if vitamin A can be supplemented at lower daily dose to malnourished children attending the Dhaka Hospital of ICDDR, B

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-59 months
2. Either sex
3. Severe malnutrition as defined by the presence of any of the followings:

   * Bipedal oedema
   * Weight (measured after correction of dehydration) for height Z score <-3 of the National Center for Health Statistics (NCHS) reference
   * Written informed consent of respective parents/ guardians for participation of the children in the study.
4. Children having diarrhoea (watery or invasive) or cough and cold or both for the last 48 hours.

Exclusion Criteria:

1. Failure to obtain consent
2. Received a dose of vitamin A within the last three months
3. History of night blindness or eye signs of vitamin A deficiency
4. Measles or history of measles within last 8 weeks [56]
5. Clinical suspicion of TB (evening rise of temperature, loss of appetite, gradual loss of weight, cough, night sweating) after applying modified Kenneth Jones criteria [57], shock other than due to hypovolaemia or hypoglycaemia, congestive cardiac failure, severe sepsis (hypothermia, tachycardia, tachypnea, hypotension) [58], and seizure disorders
6. Trisomy-21
7. Cerebral palsy
8. Any other known chronic disease (e.g. hepatic, renal or congenital disorder) or malignant condition.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260
Dates: Start 2005-10; Primary Completion 2007-12-31 (Actual); Study Completion 2007-12-31 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhoea
Resolution of ALRI

SECONDARY OUTCOMES:
Duration of acute phase of illness
Time to nutritional rehabilitation (achieving of 80% of W/H)
Rates of weight gain
Morbidity developed during hospitalization such as nosocomial infections
Measurement of Serum retinol and RBP on admission, on day 3 and on day 15
Case fatality rates

CONTACTS AND LOCATIONS:
Overall Officials: Samima Sattart, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital, ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Sattar S, Ahmed T, Rasul CH, Saha D, Salam MA, Hossain MI. Efficacy of a high-dose in addition to daily low-dose vitamin A in children suffering from severe acute malnutrition with other illnesses. PLoS One. 2012;7(3):e33112. doi: 10.1371/journal.pone.0033112. Epub 2012 Mar 27. PMID 22479361